CLINICAL TRIAL: NCT05224362
Title: Acute Effects of Elastic Band Resistance Applied to the Hip and Chest Region on Postural Stability and Physical Function Before, Immediately and up to 30 Min After Exercise in Physically Active Older Adults
Brief Title: Acute Effects of Elastic Band Resistance on Postural Stability and Physical Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Derby (Other)
Responsible Party: Principal Investigator, Nichola Davis, Principal Investigator: Miss Nichola Michelle Davis (PhD Student), University of Derby
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NDavis
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Stability; Posturography; Balance; Old Age; Debility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hip Region (Experimental): Pre intervention: Force plate Posturography Pre selected exercises (8) will be performed by the participant using an elastic resistance band anchored from ground level and placed the hip region.
  Warm up: 5-10 mins
  Exercises:
  Forward step, forward tandem steps, forward tandem hold, Upper body rotation, side steps. backward step, backward tandem walk, backward tandem hold. Cool down. Post intervention- Force plate Posturography and a Semi-structured Interview schedule
  Interventions: Device: A repeated measures acute study using using elastic resistance bands in older adults to challenge stability.
- Chest Region (Experimental): Pre intervention: Force plate Posturography Pre selected exercises (8) will be performed by the participant using an elastic resistance band anchored from ground level and placed the chest region (using velcro on a chest harness/training vest).
  Warm up: 5-10 mins
  Exercises:
  Forward step, forward tandem steps, forward tandem hold, Upper body rotation, side steps. backward step, backward tandem walk, backward tandem hold. Cool down. Post intervention- Force plate Posturography and a Semi-structured Interview schedule
  Interventions: Device: A repeated measures acute study using using elastic resistance bands in older adults to challenge stability.
- No elastic band (Placebo Comparator): Pre intervention: Force plate Posturography Pre selected exercises (8) will be performed by the participant.
  Warm up: 5-10 mins
  Exercises:
  Forward step, forward tandem steps, forward tandem hold, Upper body rotation, side steps. backward step, backward tandem walk, backward tandem hold. Cool down. Post intervention- Force plate Posturography and a Semi-structured Interview schedule
  Interventions: Device: A repeated measures acute study using using elastic resistance bands in older adults to challenge stability.

INTERVENTIONS:
Device: A repeated measures acute study using using elastic resistance bands in older adults to challenge stability. — A repeated measures acute study using using elastic resistance bands in older adults to challenge stability. Exercises with an elastic resistance band anchored from the ground and placed at the hip and chest region will be trialled. Bertec force plate analysis will be performed to assess the acute effects on balance and stability. A semi- structured interview will identify the impact and practicalities of the intervention. The information will be used in the development of an evaluation process with key consideration of the planning phase of the intervention. Questions with verbal cues to provide perceptions of the exercise selection such as likes/ dislikes, safety, confidence, difficulty, enjoyment and band placement will be asked to determine the acceptability, accessibility, appropriateness and usability of the protocol and build insights into the participant preferences.
  Other Names: Elastic Resistance Band Training; Balance training in Older Adults; Stability Training using Resistance bands in Older Adults; The acute effects of using Elastic Resistance Bands in Older Adults; Novel Elastic Resistance Band training Intervention in Older Adults; Bertec posturography; Resistance bands

SUMMARY:
Current balance and stability interventions have been shown to improve balance through targeting balance impairments and retraining effects. However, there are key facilitators and barriers 'that older adults may face to participate in such interventions'. Additionally, physical activity interventions fail to integrate older adults into the co-design and co-production of PA interventions. The study will aim to identify the impact and practicalities of an exercise intervention in older adults by performing pre selected exercises with an elastic resistance band attached at the hip and chest region to challenge balance. Static posturography will assess the impacts of the exercise intervention on balance and stability.

Researcher led interviews will focus on the participants perceptions of the activities and decision making of exercise selection by selecting components that they are confident to perform which is a key element to creating a practical and enjoyable exercise programme for the older population. This will co-create an intervention that is accessible, acceptable, and appropriate for older adults.

The study will establish the physical impact and practicalities of a novel elastic band resistance exercise intervention in older adults by performing force plate posturography and researcher led interviews that will focus on the participants perceptions of the activities and intensity levels to co-create an intervention that is accessible, acceptable, and appropriate for older adults.

DETAILED DESCRIPTION:
Outline of study designThe following study will be a repeated measures design. A convenience sample of adults/older adults will be recruited through PA networks in the Derbyshire community. Participants will not be recruited through HSN facilities or via any NHS platform. Participants will be required to attend three separate sessions with at least 48-72hours in between each session. Each session will be randomized in order to mitigate any bias and allow comparability of the 3 conditions. Experimental session one: Participants will be required to perform pre-selected exercises with an elastic resistance band placed at the hip region. Experimental session two: Participants will be required to perform pre-selected exercises with an elastic resistance band placed at the chest region. Experimental session three (control group): Participants will be required to perform pre-selected exercises without an elastic resistance band. The exercise intensity is measured throughout by RPE before, during and after each exercise.

intensity. Participants will be asked to simply perform the exercises not at any specific intensity. Force plate posturography measurements will be recorded before and immediately after and 30 minutes after the exercise intervention. The other quantitative measures (heart rate, rate of perceived exertion) will be recorded throughout the intervention and one-to-one interviews using a semi structured interview guide will be performed at the end of each session. The session order will be randomized for each participant to counterbalance the outcome which emerge from the study.

Participant preparation will include a detailed invitation to attend and briefing using a pre-prepared participant information sheet. Participants will be required to complete and return an International physical activity questionnaire, Falls efficacy scale, Confidence in maintaining balance and Instrumental Activities of Daily Living form.

Upon arrival of each session participants will be required to read and sign an informed consent form, a general health screen questionnaire and mini mental state examination. Participants will be required to complete all 3 sessions which will be supervised in the Kirtley building laboratory at the University of Derby (3 x experimental trial). Instructions will be provided for participants to abstain from alcohol and caffeine for a minimum of 12/24 hours respectively and avoidance of strenuous exercise for at least 72 hours prior to participation.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male and females over 50 years old. Although ageing is an individual and qualitative perspective rather than solely a chronological perspective, adults are transitioning to older adulthood in their 5th decade of life. Older adults may benefit from preparing at an earlier stage of ageing from the age of 50 years compared to beginning at the age of 65 years where falls are a high risk factor. PA guidelines recommend that adults will benefit from preparing physical attributes such as strength and balance at an earlier stage of the ageing process, therefore, this age group of 50 years and over has been selected as the most appropriate.
* Moderately Physically active (this will be determined by the International Physical Activity Questionnaire (IPAQ) prior to participation of the study. A score of at least 600 MET-min/week (moderate physical activity level) will be required to take part in the study.
* Ability to walk without a walking aid
* Ability to provide consent. This will be determined by using the Mini Mental State Examination (MMSE) a score of under 23. The MMSE will assess cognitive function using scoring to ensure that participants are not cognitively impaired

Exclusion Criteria:

* Individuals that are under the age of 50 years old
* Individual that have serious, unstable cardiovascular conditions such as recent acute myocardial infarction; congestive heart failure; uncontrolled hypertension; serious musculoskeletal or neurologic conditions (including Parkinson's disease, Huntington's disease, acute stroke, paresis of the lower limbs and uncontrolled diabetes mellitus.
* Individuals with acute respiratory tract infection or chronic lung disease (e.g. asthma and obstructive pulmonary disease).
* Individuals that are not physically active (METs score under 600 MET-min/ week). have severe cognitive impairment (inability to follow simple training instructions; and acute respiratory tract infection or chronic lung disease (e.g. asthma and obstructive pulmonary disease).
* Individuals that are unable to provide consent. This will be determined by using the Mini-Mental State Examination (MMSE).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Bertec Force plate posturography | through study completion, an average of 1 year
  Centre of pressure displacement and velocity parameters will be measured using a Bertec force plate and Pro-Vec software. Measurements include the position traces of anterior-posterior and mediolateral centre of pressure to provide feedback of postural stability. In particular, the mean displacement, root-mean-squared distance from mean, root-mean-square-velocity and the mean velocity of centre of pressure. Participants will stand upright and relaxed in the centre of a portable Bertec force plate with hands on hips and feet touching each other.
  Data will be collected under 4 different conditions: normal standing with eyes open, normal standing with eyes closed, a tandem stance with eyes open and a tandem stance with eyes closed. This will enable the proprioception and vestibular system to be assessed. Postural sway will be measured in the anteroposterior and mediolateral directions.
Semi structured Interview | through study completion, an average of 1 year
  A one-on-one, face to face semi-structured interview with the researcher to identify the impact and practicalities of the exercise intervention. The information will be used in the development of an evaluation process with key consideration of the planning phase of the intervention. A semi-structured interview schedule developed by the lead researcher will investigate the acceptability, accessibility, appropriateness and usability of the protocol. Participants will be asked a series of open and closed questions and likert scales to provide perceptions of the exercise selection such as likes/ dislikes, safety, confidence, difficulty, enjoyment and band placement. This will help to build insights into the participant preferences which is an important element of the intervention design.
Heart rate | through study completion, an average of 1 year
  Heart rate measures will be taken during each exercise. Higher values = higher exertion of each exercise performed. 50 beats per min - 120 = low, 120- 150 beats per min = moderate and 150 beats per min = high.
Rate of perceived exertion (RPE) | through study completion, an average of 1 year
  RPE measures will be taken during each exercise. Scale 0-10. 0= no exertion and 10 being the highest exertion exhaustion.

SECONDARY OUTCOMES:
Mini Balance Evaluation Test (MINI-BESTest) | through study completeion, an average of 1 year
  This assessment will require participants to perform a series of physical performance tasks. Following each task, the researcher will record the scores to sum a total score for the MINI BESTest. Scoring: The test has a maximum score of 28 points from 14 items that are each scored from 0-2. "0" = lowest level of function and "2" = highest level of function.
  If a subject must use an assistive device for an item, score that item one category lower.
  If a subject requires physical assistance to perform an item, score "0" for that item.
Short Falls efficacy scale (FES 1) | through study completion, an average of 1 year
  This questionnaire will require the participant to answer 7 questions on their own perceptions on concerns of falling during a series of activities. The scale for each questions is measured from a value of 1-4. 1 = not concerned at all about falling and a 4 =very concerned about falling for each item. A higher score on the FES-l will represent a greater concern for falls from a participant (lowest score 7 and highest score 28).
Balance Confidence Questionnaire (CONFbal) | through study completion, an average of 1 year
  This questionnaire contains 10 scale items which will be summed to give an index of balance confidence.

OTHER OUTCOMES:
Instrumental Activities of Daily Living form (IADL) | through study completion, an average of 1 year
  To identify how a person is functioning at the present time to determine any differences in participation recruitment. The IADL has 8 categories which the participant is required to select one out of four options that have a score assigned to their level of functioning (either 1 or 0). Scoring Interpretation: In some activities and categories, only the highest level of function receives a 1; in others, two or more levels have scores of 1 because each describes competence that represents some minimal level of function.
  These screens are useful for indicating specifically how a person is performing at the present time. Therefore a higher score on the IADL would represent a higher functioning level. Highest score= 8 (high functioning), lowest score =0 (low functioning).
International physical activity questionnaire (IPARQ) | through study completion, an average of 1 year
  IPAQ assesses physical activity undertaken across a set of domains. The following values are used for the analysis: Walking = 3.3 METs, Moderate PA = 4.0 METs and Vigorous PA = 8.0 METs. Low= Individuals who not meet criteria for Categories 2 or 3 are considered to have a 'low' physical activity level. Moderate= a) 3 or more days of vigorous-intensity activity of at least 20 minutes per day b) 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day c) 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum Total physical activity of at least 600 MET-minutes/week. High= a) vigorous-intensity activity on at least 3 days achieving a minimum Total physical activity of at least 1500 MET minutes/week b) 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum Total physical activity of at least 3000 MET-minutes/week.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Pringle, Study Director — University of Derby
Locations (2):
- United Kingdom (2):
  - University of Derby, Derby
  - University Of Derby, Derby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barry BK, Carson RG. The consequences of resistance training for movement control in older adults. J Gerontol A Biol Sci Med Sci. 2004 Jul;59(7):730-54. doi: 10.1093/gerona/59.7.m730. PMID 15304540
- [Result] Carroll TJ, Barry B, Riek S, Carson RG. Resistance training enhances the stability of sensorimotor coordination. Proc Biol Sci. 2001 Feb 7;268(1464):221-7. doi: 10.1098/rspb.2000.1356. PMID 11217890
- [Result] Colado JC, Garcia-Masso X, Pellicer M, Alakhdar Y, Benavent J, Cabeza-Ruiz R. A comparison of elastic tubing and isotonic resistance exercises. Int J Sports Med. 2010 Nov;31(11):810-7. doi: 10.1055/s-0030-1262808. Epub 2010 Aug 11. PMID 20703977
- [Result] Colado JC, Triplett NT. Effects of a short-term resistance program using elastic bands versus weight machines for sedentary middle-aged women. J Strength Cond Res. 2008 Sep;22(5):1441-8. doi: 10.1519/JSC.0b013e31817ae67a. PMID 18714245
- [Result] Gardner MM, Buchner DM, Robertson MC, Campbell AJ. Practical implementation of an exercise-based falls prevention programme. Age Ageing. 2001 Jan;30(1):77-83. doi: 10.1093/ageing/30.1.77. PMID 11322678
- [Result] Gerards MHG, McCrum C, Mansfield A, Meijer K. Perturbation-based balance training for falls reduction among older adults: Current evidence and implications for clinical practice. Geriatr Gerontol Int. 2017 Dec;17(12):2294-2303. doi: 10.1111/ggi.13082. Epub 2017 Jun 16. PMID 28621015
- [Result] Lima FF, Camillo CA, Gobbo LA, Trevisan IB, Nascimento WBBM, Silva BSA, Lima MCS, Ramos D, Ramos EMC. Resistance Training using Low Cost Elastic Tubing is Equally Effective to Conventional Weight Machines in Middle-Aged to Older Healthy Adults: A Quasi-Randomized Controlled Clinical Trial. J Sports Sci Med. 2018 Mar 1;17(1):153-160. eCollection 2018 Mar. PMID 29535589
- [Result] Mansfield A, Aqui A, Centen A, Danells CJ, DePaul VG, Knorr S, Schinkel-Ivy A, Brooks D, Inness EL, McIlroy WE, Mochizuki G. Perturbation training to promote safe independent mobility post-stroke: study protocol for a randomized controlled trial. BMC Neurol. 2015 Jun 6;15:87. doi: 10.1186/s12883-015-0347-8. PMID 26048054
- [Result] Mansfield A, Peters AL, Liu BA, Maki BE. A perturbation-based balance training program for older adults: study protocol for a randomised controlled trial. BMC Geriatr. 2007 May 31;7:12. doi: 10.1186/1471-2318-7-12. PMID 17540020
- [Result] Youdas JW, Adams KE, Bertucci JE, Brooks KJ, Nelson MM, Hollman JH. Muscle activation levels of the gluteus maximus and medius during standing hip-joint strengthening exercises using elastic-tubing resistance. J Sport Rehabil. 2014 Feb;23(1):1-11. doi: 10.1123/jsr.2012-0082. Epub 2013 Aug 6. PMID 23921445
- See also: NHS balance exercises — https://www.nhs.uk/live-well/exercise/balance-exercises/
- See also: NHS Overview on Falls — https://www.nhs.uk/conditions/Falls/
- See also: Department of Health Older Adults Physical Activity Guidelines — https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/832868/uk-chief-medical-officers-physical-activity-guidelines.pdf
- See also: National falls and fracture prevention strategy 2019-2024 — https://www.gov.scot/publications/national-falls-fracture-prevention-strategy-scotland-2019-2024/pages/7/